CLINICAL TRIAL: NCT01455623
Title: Development and Validation of a Disability Severity Index for Charcot Marie Tooth Disease
Brief Title: Development and Validation of a Disability Severity Index for CMT
Acronym: 6604
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Muscular Dystrophy Association (Other)
Responsible Party: Principal Investigator, Michael Shy, Professor, University of Iowa
Other Study IDs: INC-6604
Record Dates: First submitted 2011-10-17; First posted 2011-10-20 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Charcot Marie Tooth Disease
Keywords: CMT
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Health Care Provider: A person working within the field of CMT.
- Patient with CMT: Any person of any age self-identifying as having CMT and belonging to the Inherited Neuropathies Consortium Contact Registry hosted by the Rare Disease Clinical Research Network.

SUMMARY:
It is necessary for outcome measures to accurately reflect the state of health of a person in order for clinical trials to show benefit. The most commonly used outcome measure for Charcot Marie Tooth Disease (CMT) is the CMT Neuropathy Score, which uses cutoffs of points designated as mild (0-10 points), moderate (11-20) or severe (21-36). These terms are arbitrary. This study is looking to base mild, moderate, and severe on what both people affected with CMT and those who provide for people with CMT consider appropriate.

ELIGIBILITY:
Inclusion Criteria:

* patients with CMT ages 8-100,
* health care professionals who take care of patients with CMT.

  * Eligible patients will be patients that have joined the INC RDCRN Contact Registry. These will be patients or guardians with known or probable inherited neuropathies.
  * Eligible health care professionals who participate in the care of patients with inherited neuropathies (physicians, genetic counselors, physical and occupational therapists etc.) attending the 4th International CMT Consortium to be held in Potomac Maryland June 29-July 1, 2011.

Exclusion Criteria:

* Does not read or speak English.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Two cohorts:
  1. Patients self identified as having CMT and have chosen to be a part of the Inherited Neuropathies Consortium Contact Registry, housed by the Rare Disease Clinical Research Network.
  2. Healthcare Providers working in the field of CMT.
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2011-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Compare Patient and Healthcare Provider impressions of what constitutes mild, moderate and severe impairment in CMT | 1 year

SECONDARY OUTCOMES:
Develop a Disability Severity Index including items with high patient-physician concordance | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sindhu Ramchandren, MD, Principal Investigator — Wayne State University
Locations (1):
- University of Iowa, Iowa City, Iowa, United States